CLINICAL TRIAL: NCT00992654
Title: A Local, Multicentre, Open Label Access Program To Provide Maraviroc To Eligible Adult Patients Completing A4001050 Study Until Commercial Availability Of Maraviroc (Celsentri) In India
Brief Title: A Treatment Access Program To Provide Maraviroc To Eligible Adult Patients Completing A4001050 Study Until Commercial Availability Of Maraviroc (Celsentri) In India
Status: No longer available | Type: Expanded Access
Sponsor: ViiV Healthcare (Industry)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: A4001096; A4001050
Record Dates: First submitted 2009-10-08; First posted 2009-10-09 (Estimated); Last update posted 2018-09-27 (Actual); Status verified 2018-09

CONDITIONS: Human Immunodeficiency Virus (HIV)
Keywords: Open Label Access Program; Treatment experienced
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — Maraviroc

INTERVENTIONS:
Drug: Open Label Treatment Access: Maraviroc — Oral dosing twice daily. The dose will depend on the optimized background therapy.
  Other Names: Maraviroc, Celsentri, Selzentry

SUMMARY:
The new protocol will allow the patients enrolled on A4001050 to have continuous access of Maraviroc and the treatment will not be interrupted until the drug is commercially available in India.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who complete the A4001050 study and are continuing to derive benefit from Maraviroc.
* Subjects who are willing and able to comply with scheduled visits, treatment plan and other study procedures.

Exclusion Criteria:

* Subjects who discontinued in A4001050 study.
* Unable to provide consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A4001096&StudyName=A%20Treatment%20Access%20Program%20To%20Provide%20Maraviroc%20To%20Eligible%20Adult%20Patients%20Completing%20A4001050%20Study%20Until%20Commercial%20Availability%20Of%20Mara